CLINICAL TRIAL: NCT01618474
Title: A Phase II Randomized Controlled Trial of Adjuvant Chemotherapy for High Risk Gastric Cancer Patients (IIIb-IIIc)
Brief Title: Trial of Adjuvant Chemotherapy for High Risk Gastric Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIH-HDZ-201205001
Record Dates: First submitted 2012-05-27; First posted 2012-06-13 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-05

CONDITIONS: Stomach Cancer
Keywords: gastric cancer; adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Capecitabine; XELOX; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DX (Experimental): DX: Docetaxel 60mg/m2, intravenous infusion, day 1; Capecitabine 1000mg/m2, oral administration, twice a day, day1-14; 3 weeks a cycle for 8 consecutive cycles.
  Interventions: Drug: DX
- XELOX (Active Comparator): XELOX: oxaliplatin 130mg/m2, intravenous infusion, day 1; Capecitabine 1000mg/m2, oral administration, twice a day, day 1-14, 3 weeks a cycle for 8 consecutive cycles
  Interventions: Drug: XELOX

INTERVENTIONS:
Drug: DX — Docetaxel 60mg/m2, intravenous infusion, day 1; Capecitabine 1000mg/m2, oral administration, twice a day, day1-14; 3 weeks a cycle for 8 consecutive cycles.
  Other Names: Docetaxel; Xeloda
  Arms: DX
Drug: XELOX — oxaliplatin 130mg/m2, intravenous infusion, day 1; Capecitabine 1000mg/m2, oral administration, twice a day, day 1-14, 3 weeks a cycle for 8 consecutive cycles
  Other Names: Eloxatin; XEloda
  Arms: XELOX

SUMMARY:
This trial is going to evaluate the efficacy and safety of two regimens of DX (docetaxel plus capecitabine)and XELOX (oxaliplatin plus capecitabine)as adjuvant chemotherapy for stage IIIb-IIIc gastric cancer patients after curative D2/D2+ operation, and to investigate the optimal adjuvant regimen for such extremely high risk patients.

DETAILED DESCRIPTION:
Operation is the only curative treatment for gastric cancer patients. However, the rate of recurrence is high up to 60%. The 5 year's overall survival of patient at stage IIIb or more advanced stage is still poor and approximately 8-28%. Adjuvant chemotherapy is critical for improving efficacy further. Unfortunately, the optimal adjuvant regimen is not identified yet. The standard adjuvant treatments of American and European patients are not accepted widely in Asia area because of different operation procedure and patient's tolerability. Results of two critical trials indicated that S-1 alone as Japanese standard adjuvant chemotherapy could not improve the survival of stage IIIb advanced stage gastric cancer patients while the Korean standard regimen XELOX could. This implied that the more intensive chemotherapy must be used for the patients with higher risk of relapse. The proportion of the stage IIIb-IIIc Chinese gastric cancer patients is much larger than that of Japan and Korean. However, no randomized trial focusing on the extremely high risk of relapse stage IIIb and stage IIIc patients has been performed, and the standard adjuvant chemotherapy regimen is not clear and needs to be investigated.

Docetaxel based combination is one of the most effective regimens for advanced gastric cancer. The combination of docetaxel and 5-FU was found to have a similar efficacy to ECF regimen along with milder toxicity. Capecitabine has been proved to be a good alternative to infusional 5-FU. So, docetaxel plus capecitabine seems to be a promising adjuvant regimen for high risk stage IIIb-IIIc gastric cancer patients. But it still needs to be verified.

This trial is going to evaluate the efficacy and safety of two regimens of DX and XELOX as adjuvant chemotherapy for stage IIIb-IIIc gastric cancer patients after curative D2/D2+ operation, and to investigate the optimal adjuvant regimen for such extremely high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* a post operation histologically confirmed gastric or esophagogastric junction adenocarcinoma;
* curative D2 or D2+ operation had been performed, and the pathological stage post operation was verified as IIIb or IIIc;
* no adjuvant chemotherapy before or after operation;
* Karnofsky performance status scale ≥ 70;
* prior adjuvant chemotherapy that did not include taxanes and S-1;
* white blood count ≥ 3,500/mm3, absolute neutrophil count ≥ 1,500/mm3, platelet count ≥ 100,000/mm3, hemoglobin count ≥ 90 g/dL, serum bilirubin level < 1.5 of the upper limit of normal (ULN) for the institution, aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase ≤ 2.5 ULN, serum albumin ≥ 30g/L, serum creatinine ≤ 1.5 ULN; and
* normal cardiac function with no severe heart disease.

Exclusion Criteria:

Major exclusion criteria were as follows:

* pregnancy or breast feeding;
* past history of allergy to taxanes, platinum and 5-fluorouracil or their analogues;
* radiotherapy for all measurable target lesions;
* obstructive bowel disease;
* past history of other cancers except for cured non-melanoma skin cancer or cervical cancer; and
* concomitant treatment with other anticancer drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years
  DFS was difined as the length of time from the date of randomization to the date of first documentation of relapse of gastric cancer or any other type of cancer or death.

SECONDARY OUTCOMES:
overall survival | 3 years
  OS was defined as the length of time from the date of randomization to the date of death of vaious reasons
CTC negative conversion rate | 3 years
  CTC negative conversion rate was defined as the proportion of the patients whose positive circulating tumor cell turns to be negative after adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, M.D., Principal Investigator — Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China